CLINICAL TRIAL: NCT02598856
Title: Bioavailability of Nasal Naloxone and Injected Naloxone Compared. A Randomized, Open Label, 4-way Cross-over Study
Brief Title: Bioavailability of Nasal Naloxone and Injected Naloxone Compared
Acronym: OPI-15-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); A/S Den norske Eterfabrikk (Industry); Smerud Medical Research International AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OPI 15-002; 2015-002355-10 (EudraCT Number)
Record Dates: First submitted 2015-11-02; First posted 2015-11-06 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Drug Overdose
Keywords: Emergency Treatment; Morphine Derivates; Heroin; Antidotes; Administration, Intravenous; Pharmacology; Naloxone; Healthy volunteers; Administration, intramuscular; Administration, intranasal
MeSH Terms: conditions — Drug Overdose | interventions — Naloxone; Injections, Intramuscular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Intranasal naloxone 1x (Experimental): Each subject will receive one dose of IN naloxone 1.4 mg, IN naloxone 2 x 1.4 mg, IV naloxone 0.4 mg and IM naloxone 0.8 mg in a randomized order. The four doses will be given at four different visits with a washout period of at least 72 hours between. One follow-up visit will be conducted within one month after the last exposure.
  Interventions: Drug: Intranasal (IN) naloxone 1x; Drug: Intranasal (IN) naloxone 2; Drug: Intravenous (IV) naloxone; Drug: Intramuscular (IM) naloxone
- Intranasal naloxone 2x (Active Comparator): Each subject will receive one dose of IN naloxone 1.4 mg, IN naloxone 2 x 1.4 mg, IV naloxone 0.4 mg and IM naloxone 0.8 mg in a randomized order. The four doses will be given at four different visits with a washout period of at least 72 hours between. One follow-up visit will be conducted within one month after the last exposure.
  Interventions: Drug: Intranasal (IN) naloxone 1x; Drug: Intranasal (IN) naloxone 2; Drug: Intravenous (IV) naloxone; Drug: Intramuscular (IM) naloxone
- Intravenous naloxone (Active Comparator): Each subject will receive one dose of IN naloxone 1.4 mg, IN naloxone 2 x 1.4 mg, IV naloxone 0.4 mg and IM naloxone 0.8 mg in a randomized order. The four doses will be given at four different visits with a washout period of at least 72 hours between. One follow-up visit will be conducted within one month after the last exposure.
  Interventions: Drug: Intranasal (IN) naloxone 1x; Drug: Intranasal (IN) naloxone 2; Drug: Intravenous (IV) naloxone; Drug: Intramuscular (IM) naloxone
- Intramuscular naloxone (Active Comparator): Each subject will receive one dose of IN naloxone 1.4 mg, IN naloxone 2 x 1.4 mg, IV naloxone 0.4 mg and IM naloxone 0.8 mg in a randomized order. The four doses will be given at four different visits with a washout period of at least 72 hours between. One follow-up visit will be conducted within one month after the last exposure.
  Interventions: Drug: Intranasal (IN) naloxone 1x; Drug: Intranasal (IN) naloxone 2; Drug: Intravenous (IV) naloxone; Drug: Intramuscular (IM) naloxone

INTERVENTIONS:
Drug: Intranasal (IN) naloxone 1x — Administered as 100 μl 14.0 mg/ml (1.4 mg naloxone) by Aptar Unitdose device as one puff in one nostril
Drug: Intranasal (IN) naloxone 2 — Administered as 2x 100 μl 14 mg/ml (2.8 mg naloxone) by Aptar Unitdose device as two puffs within the same nostril with 3 minutes interval
Drug: Intravenous (IV) naloxone — Administered as 1 ml Naloxon B Braun 0.4 mg/ml (0.4 mg naloxone), in an intravenous cannula in the opposite arm of which the blood samples are drawn from. IV bolus will be given rapidly (in less than 5 seconds)
Drug: Intramuscular (IM) naloxone — Naloxone administered as 2 ml Naloxon B Braun 0.4 mg/ml (0.8 mg naloxone) in a Braun Omnifix 2.5 ml syringe using a BD Microlance 3 21G (green) 0.8x40 mm needle in the deltoid muscle of the non-dominant arm

SUMMARY:
Opioid overdoses have in the last decade counted for about 230 untimely deaths annually in Norway. The government is currently implementing a strategy for combating this epidemic. Among the actions promoted in this strategy is the distribution of naloxone for intranasal administration. Such administration of naloxone is currently being implemented and tried out around the world, but very little has been done to pharmacologically study this new route of administration of this well known drug, and only 3 open label randomized controlled trials (RCTs) have been conducted. A recent guideline from the WHO on community management of opioid overdoses is a comprehensive review of many of the aspects the investigators cover in our research.

Regarding both dosage, routes of administration of naloxone and care of these patients in the pre hospital setting. The WHO calls for nasal formulations with a higher concentration, as well as focuses on the current wide spread off label use of nasal naloxone as a problem and identifies several research questions of critical importance and very low evidence.The current study, together with our research group's previous and future studies, aims to provide data for the development of a medicinal product with marketing authorisation for use in pre-hospital overdoses. This to contribute to public health measures for opioid users and those around them.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study the subjects must meet all of the following inclusion criteria:

* Provision of a signed written informed consent
* ECG without any pathological abnormalities
* Have a BMI range of 18.5- 26.0 kg/m
* Female subject with child bearing potential must use high efficacy contraception. For the purpose of this study acceptable contraception is defined as sterilization, oral contraceptives, patch, implants, vaginal ring, hormonal IUD or copper IUD through out the study until the last visit.
* Laboratory values within reference values for the following haematology and biochemistry tests:

  * Haemoglobin
  * Creatinine
  * ASAT
  * ALAT
  * Gamma GT

Exclusion Criteria:

In order to participate in the study subjects must not meet any of the following exclusion criteria:

* using medication on a regular basis, including regular use of nasal spray of any form.
* History of prior drug allergy
* local nasal disease or nasal surgery for the last 2 months
* Pregnant or breast feeding women. A serum HCG below 3 U/L must be demonstrated in females of child-bearing potential at Screening Visit.
* Current drug or alcohol abuse, which in the opinion of the Investigator should preclude participation in the study.
* Having received another new medical chemical entity (defined as a compound which has not been approved for marketing) or having participated in any other clinical study that included drug treatment within 3 months of the administration of investigational product in this study.
* Hypersensitivity to naloxone or any of its excipients.
* Investigator considers subject unlikely to comply with study procedures, restrictions and/or other requirements.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Difference in Peak plasma concentration (Cmax) | 4 days
  Cmax will be compared for single dose IN, IM and IV naloxone
Difference in systemic exposure: Area under the plasma concentration versus time curve (AUC-0last) | 4 days
  AUC 0-last will be compared for single dose IN, IM and IV naloxone
Difference in dose adjusted systemic exposure: Area under the plasma concentration versus time curve (AUC-0inf) | 4 days
  AUC0-inf will be compared for single dose IN, IM and IV naloxone
Difference in time at which the Cmax is observed (Tmax) | 4 days
  Tmax will be compared for single dose IN, IM and IV naloxone

SECONDARY OUTCOMES:
Dose proportionality | 4 days
  assessed by comparing systemic exposure (AUC0-last) following one and two doses of 1.4 mg of IN naloxone in the same nostril.
Absolute bioavailability | 4 days
  assessed by comparing dose adjusted systemic exposure (AUC0-last) of IN and IV naloxone
Relative bioavailability | 4 days
  assessed by comparing dose adjusted systemic exposure (AUC0-last) of IN and IM naloxone

CONTACTS AND LOCATIONS:
Overall Officials: Toril A Nagelhus Hernes, phd prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway